CLINICAL TRIAL: NCT02210247
Title: An Open-Label Cohort Study to Evaluate the Safety and Pharmacokinetics of Redosing EXPAREL Via Local Subcutaneous Infiltration in Healthy Volunteers
Brief Title: Safety and Pharmacokinetics Study of Redosing EXPAREL in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 402-C-113
Record Dates: First submitted 2014-08-04; First posted 2014-08-06 (Estimated); Results first posted 2021-07-02 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Active Comparator): Cohort 1 will receive a single dose of EXPAREL 266 mg on Day 1. No additional dose will be given.
  Interventions: Drug: EXPAREL
- Cohort 2 (Active Comparator): Cohort 2 will receive a dose of EXPAREL 266 mg on Day 1 and a second dose of EXPAREL 266 mg on Day 4 at 72 hours.
  Interventions: Drug: EXPAREL
- Cohort 3 (Active Comparator): Cohort 3 will receive a dose of EXPAREL 266 mg on Day 1 and a second dose of EXPAREL 266 mg on Day 3 at 48 hours.
  Interventions: Drug: EXPAREL
- Cohort 4 (Active Comparator): Cohort 4 will receive a dose of EXPAREL 266 mg on Day 1 and a second dose of EXPAREL 266 mg on Day 2 at 24 hours.
  Interventions: Drug: EXPAREL
- Cohort 5 (Active Comparator): Cohort 5 will receive a single dose of EXPAREL 266 mg on Day 1 followed immediately by a second dose of EXPAREL 266 mg (total of 532 mg/40 mL).
  Interventions: Drug: EXPAREL

INTERVENTIONS:
Drug: EXPAREL
  Other Names: bupivacaine liposome injectable suspension

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics of redosing EXPAREL via local subcutaneous infiltration in healthy volunteers.

DETAILED DESCRIPTION:
During Dosing Period 1, blood samples for pharmacokinetic (PK) analysis will be obtained predose (15 minutes prior to administration of EXPAREL) through 12 hours postdose (i.e., at 15 and 30 minutes, 1, 2, 4, 8, and 12 hours) for Cohort 4; through 36 hours postdose (i.e., at 15 and 30 minutes, 1, 2, 4, 8, 12, 24, and 36 hours) for Cohort 3; through 60 hours postdose (i.e., at 15 and 30 minutes, 1, 2, 4, 8, 12, 24, 36, 48, and 60 hours) for Cohort 2; and through 72 hours postdose (i.e., at 15 and 30 minutes, 1, 2, 4, 8, 12, 24, 36, 48, 60, and 72 hours) for Cohorts 1 and 5.

During Dosing Period 2 (Cohorts 2, 3, and 4 only), blood samples for PK analysis will be obtained predose (15 minutes prior to administration of EXPAREL) through 72 hours postdose (i.e., at 15 and 30 minutes, 1, 2, 4, 8, 12, 24, 36, 48, 60, and 72 hours).

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥18 years of age.
* American Society of Anesthesiologists (ASA) physical status 1 or 2.
* Female subjects must be surgically sterile, at least 2 years postmenopausal, or using a medically acceptable method of birth control. If of childbearing potential, must have a documented negative pregnancy test within 24 hours before the first study drug administration.
* Able to provide informed consent, adhere to the study visit schedule, and complete all study assessments.

Exclusion Criteria:

* History of hypersensitivity or idiosyncratic reactions to amide-type local anesthetics.
* History of abnormal bleeding tendencies/clotting disorders.
* Regular use of anticoagulants (except for low dose aspirin for cardioprotection).
* Received any investigational drug within 30 days prior to study drug administration, and/or has planned administration of another investigational product or procedure during his/her participation in this study.
* Currently pregnant, nursing, or planning to become pregnant during the study or within 1 month after study drug administration.
* Subjects with significant medical conditions or laboratory results that, in the opinion of the Investigator, would constitute a contraindication to participation in the study, or cause inability to comply with the study requirements.
* Received bupivacaine or other local anesthetic within 7 days of first study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Biernat, MD, Principal Investigator — Medpace Clinical Pharmacology Unit
Locations (1):
- Medpace Clinical Pharmacology Unit, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Rice D, Heil JW, Biernat L. Pharmacokinetic Profile and Tolerability of Liposomal Bupivacaine Following a Repeated Dose via Local Subcutaneous Infiltration in Healthy Volunteers. Clin Drug Investig. 2017 Mar;37(3):249-257. doi: 10.1007/s40261-017-0495-2. PMID 28120158

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Cohort 1 received a single dose of EXPAREL 266 mg on Day 1. No additional dose was given.
  EXPAREL
- Cohort 2: Cohort 2 received a dose of EXPAREL 266 mg on Day 1 and a second dose of EXPAREL 266 mg on Day 4 at 72 hours.
  EXPAREL
- Cohort 3: Cohort 3 received a dose of EXPAREL 266 mg on Day 1 and a second dose of EXPAREL 266 mg on Day 3 at 48 hours.
  EXPAREL
- Cohort 4: Cohort 4 received a dose of EXPAREL 266 mg on Day 1 and a second dose of EXPAREL 266 mg on Day 2 at 24 hours.
  EXPAREL
- Cohort 5: Cohort 5 received a single dose of EXPAREL 266 mg on Day 1 followed immediately by a second dose of EXPAREL 266 mg (total of 532 mg/40 mL).
  EXPAREL
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Started | 12 | 12 | 12 | 12 | 12
Completed | 12 | 12 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (11.90) | 37.8 (11.66) | 36.9 (10.83) | 41.6 (12.38) | 44.1 (14.56) | 41.2 (12.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 0 | 2 | 8 | 6 | 23
  Male | 5 | 12 | 10 | 4 | 6 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 12 | 12 | 12 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 10 | 9 | 9 | 8 | 42
  White | 6 | 2 | 3 | 3 | 4 | 18
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 12 | 12 | 60

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Time Frame: Period(P)1 all cohorts (C) 15 m in pre, 15,30m, 1,2,34,8,12h postdose. C3: +24, 36 h postdose. C2: C3+48,60h postdose; C1 and C5: C2+72h postdose; P2: C2,3,4 only: 15m pre, 1,2,4,8,12,24,36,48,60,72h postdose. Final at D14- all subjects
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cohort 1: Cohort 1 will receive a single dose of EXPAREL 266 mg on Day 1. No additional dose will be given.
  EXPAREL
- Cohort 2: Cohort 2 will receive a dose of EXPAREL 266 mg on Day 1 and a second dose of EXPAREL 266 mg on Day 4 at 72 hours.
  EXPAREL
- Cohort 3: Cohort 3 will receive a dose of EXPAREL 266 mg on Day 1 and a second dose of EXPAREL 266 mg on Day 3 at 48 hours.
  EXPAREL
- Cohort 4: Cohort 4 will receive a dose of EXPAREL 266 mg on Day 1 and a second dose of EXPAREL 266 mg on Day 2 at 24 hours.
  EXPAREL
- Cohort 5: Cohort 5 will receive a single dose of EXPAREL 266 mg on Day 1 followed immediately by a second dose of EXPAREL 266 mg (total of 532 mg/40 mL).
  EXPAREL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
ng/mL | 129 (47) | 207 (57) | 202 (74) | 290 (119) | 246 (78)

2. Primary Outcome: Time to Maximum Concentration (Tmax)
Time Frame: Period(P)1 all cohorts 15 m in pre, 15,30m, 1,2,34,8,12h postdose. C3: +24, 36 h postdose. C2: C3+48,60h postdose; C1 and C5: C2+72h postdose; P2: C2,3,4 only: 15m pre, 1,2,4,8,12,24,36,48,60,72h postdose. Final at D14- all subjects
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
hours | 24 [24 to 72] | 48 [24 to 72] | 48 [1 to 72] | 36 [24 to 72] | 24 [8 to 72]

3. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time 0 to the Time of the Last Quantifiable Concentration [AUC(0-last)]
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: H*ng/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
H*ng/mL | 5917 (1738) | 10976 (2879) | 10201 (3721) | 15227 (7463) | 11567 (3737)

4. Primary Outcome: Apparent Terminal Elimination Half-life
Time Frame: as for outcome 2
Population: Where n per group <12, values were either not calculated or not reported.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 2 | 6 | 6 | 2 | 7
hours | 80.24 (22.64) | 44.88 (25.64) | 51.70 (26.99) | 33.22 (3.80) | 59.13 (25.03)

5. Primary Outcome: The Apparent Terminal Elimination Rate Constant (λz)
Time Frame: as for outcome 2
Population: Where n per group <12, values were either not calculated or not reported.
Measure: Mean (Standard Deviation); unit: 1/hours
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 2 | 6 | 6 | 2 | 7
1/hours | 0.009 (0.003) | 0.019 (0.007) | 0.016 (0.007) | 0.021 (0.002) | 0.014 (0.006)

ADVERSE EVENTS:
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 5/12 | 2/12 | 7/12 | 2/12 | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=12) | Cohort 2 (N=12) | Cohort 3 (N=12) | Cohort 4 (N=12) | Cohort 5 (N=12)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection-site reaction (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Vessel puncture site haematoma (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No